CLINICAL TRIAL: NCT02148133
Title: A Non-randomized, Open-label, Phase II Study to Assess the Safety and Efficacy of Eltrombopag in Japanese Subjects With Refractory, Moderate or More Severe Aplastic Anemia
Brief Title: A Study to Assess the Safety and Efficacy of Eltrombopag in Japanese Subjects With Refractory, Moderate or More Severe Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200926; CETB115E1201 (Other: Novartis)
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-01

CONDITIONS: Cytopaenia
Keywords: Eltrombopag; Aplastic Anemia (AA); Thrombocytopenia; Thrombopoietin; Bone Marrow; Bone Marrow Biopsy; Hematopoietic Stem Cells; Mature Blood Cells; Pancytopenia; Leukopenia; Platelets
MeSH Terms: conditions — Anemia, Aplastic; Thrombocytopenia; Jacobs syndrome; Pancytopenia; Leukopenia | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eltrombopag (Experimental): Subjects were assigned the investigational product (eltrombopag 25 mg/day) orally once a day under fasting condition. The dose adjustment was done every 2 weeks according to the platelet count (increased by eltrombopag 25 mg/day every 2 weeks according to the platelet count up to 100 mg/day).
  Interventions: Drug: Eltrombopag 12.5 mg; Drug: Eltrombopag 25 mg

INTERVENTIONS:
Drug: Eltrombopag 12.5 mg — White, round, film-coated tablets containing 12.5 mg of eltrombopag free acid (SB-497115-GR, eltrombopag) in each tablet
  Other Names: Revolade
Drug: Eltrombopag 25 mg — White, round, film-coated tablets containing 25 mg of eltrombopag free acid (SB-497115-GR, eltrombopag) in each tablet
  Other Names: Revolade

SUMMARY:
This was a non-randomized, open-label, phase II study to assess the efficacy and safety of eltrombopag in Japanese moderate or more severe aplastic anemia (AA) subjects with a platelet count <30,000/microliter who were refractory to anti-thymocyte globulin (ATG)-based immunosuppressive therapy (IST), who have relapsed after ATG-based IST, or who are ineligible for ATG-based IST.

Eltrombopag was expected to improve trilineage blood cells and decrease transfusion frequency based on the result from the previous study in patients with severe AA. This study used the hematologic response rate, defined as the proportion of subjects showing improvement in at least one of the three blood cell lineages or a decrease in blood transfusion volume, as the primary endpoint.

A total of 36 subjects were screened and 21 were enrolled in the study. Treatment with eltrombopag started at 25 milligram (mg)/day and increased by 25 mg/day every 2 weeks according to the platelet count up to 100 mg/day. Response assessment was performed at 3 months after starting the study treatment (Week 13). Subjects in whom the treatment was assessed as effective continued with the study treatment. Subjects in whom the treatment was assessed as effective (when meeting any of the response criteria) at 6 months after starting the study treatment (Week 26) might enter the extension phase and continue the treatment with eltrombopag. The primary endpoint was the hematologic response rate at Week26.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject has given written informed consent. If a subject is under 20 years, both the subject and the subject's legally acceptable representative have to give informed consent.
* Japanese subjects aged >=18 and <80 years at the time of informed consent.
* Diagnosis of moderate (stage II) or more Aplastic Anemia (AA) with platelet count <30,000/microliter (based on the diagnosis criteria of AA established by the Study Group on Idiopathic Hematopoietic Disorder as a part of Research on Measures for Intractable Diseases supported by Health and Labor Science Research Grants).
* Subjects who became refractory to Anti-thymocyte globulin (ATG)-based Immunosuppressive therapy (IST), who have relapsed after ATG-based IST, or who are ineligible for ATG-based IST. Note: Refractory or relapsed subjects to whom re-treatment with ATG is indicated should not be enrolled in the study. Subjects who have a sibling donor with matched human leukocyte antigen (HLA) should not be enrolled in the study. However, such subjects may be enrolled if the disease relapsed after hematopoietic stem cell transplantation (HSCT), if HSCT is not indicated, or the subject does not want to undergo HSCT.
* Adequate organ function at screening and Day 1 as defined as follows: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=3 × central laboratory upper limit of normal (ULN); Creatinine, total bilirubin, and alkaline phosphatase (ALP) <1.5 × central laboratory ULN (total bilirubin <2.5 × central laboratory ULN with Gilbert's Syndrome)
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS): 0 or 1
* Subjects with QT interval corrected for heart rate by Fridericia's formula (QTcF) <450 milliseconds (msec) or QTcF<480 msec with branch block. Corrected QT interval duration (QTc) is QT interval corrected by Fridericia formula (QTcF), machine or manual over read. QTcF is based on single or averaged QTc value of triplicate electrocardiogram (ECG).
* Subjects who meet one of the following conditions: Male subjects who have a female partner of childbearing potential must either have a prior vasectomy or agree to use an acceptable contraception from time of enrollment in the study until 16 weeks after the last dose of eltrombopag (based upon the lifecycle of sperm); Female subjects of non-childbearing potential (who are physiologically unable to become pregnant) defined as: Premenopausal women with documented bilateral oophorectomy, bilateral tubal ligation, or hysterectomy; or postmenopausal women after at least 12 months of natural amenorrhea [if uncertain, postmenopausal state should be confirmed by hematology result of follicle stimulating hormone (FSH) >40 milli international unit /milliliter (mIU/mL) or estradiol <40 picogram (pg)/mL (<140 picomole /Liter (pmole/L)].; Female subjects of childbearing potential: Defined as those not meeting the definition of non-childbearing potential. Female subjects of childbearing potential must have a negative serum human chorionic gonadotropin (hCG) or urine pregnancy test within 7 days prior to the first dose of study treatment. It is recommended that the pregnancy test should be performed as close as possible to the first dose of study treatment. Female subjects with a positive pregnancy test must be excluded from the study. Subjects with a negative pregnancy test must use acceptable contraception including abstinence after the pregnancy test. Subjects must agree to use the acceptable contraception including abstinence from 14 days prior to the first dose of study treatment until 28 days after the last dose of eltrombopag.

Key Exclusion Criteria:

* Treatment with ATG in the past 12 months. Note: Subjects who are receiving cyclosporine or anabolic steroids (excluding danazol) at a stable dose may be enrolled if laboratory values are stable at screening.
* Congenital aplastic anemia (e.g., Fanconi anemia, congenital dyskeratosis)
* Paroxysmal nocturnal hemoglobinuria (PNH) granulocyte clone size determined by flow cytometry >=50%
* Presence of chromosomal aberration (-7/7q- detected by fluorescence in situ hybridization (FISH), or other aberrations detected by Giemsa (G)-band staining) Note: Subjects with the result by G-band staining (bone marrow aspiration) not adopted into the abnormal clone definition of An International System for Human Cytogenetic Nomenclature (ISCN) can be enrolled as no chromosomal aberration.
* Past history of thromboembolism or current use of anticoagulants. Note: Subjects with antiphospholipid antibody syndrome (APS) should not be enrolled.
* Past or current history of malignant tumor. Note: Subjects who have a history of completely resected malignant tumor and have been disease-free for 5 years are eligible.
* Subjects who test positive for hepatitis B surface (HBs) antigen, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody at screening. Note: Subjects with inactive hepatitis B may be enrolled. Judgment of inactive hepatitis B will be done by the medical advisor.
* Subjects with concurrent uncontrollable severe infection (e.g., sepsis)
* Hepatic cirrhosis
* Cardiac disorder (congestive heart disease of New York Heart Association (NYHA) functional classification Grade II/III/IV), or arrhythmia with a risk of thrombosis (e.g., atrial fibrillation). Note: Subjects with NYHA Grade II due to cardiac disorder should not be enrolled but those with NYHA Grade II due to Aplastic Anemia (AA) may be enrolled.
* Alcohol or drug abuse
* Pregnant women (a positive serum or urine pregnancy test within 7 days prior to the first dose of study treatment) or lactating women. Note: Female subjects who are lactating are eligible to participate if they discontinue nursing prior to the first dose of study treatment and refrain from nursing until 5 days after the treatment completion.
* Past history of immediate or delayed hypersensitivity to compounds chemically similar to eltrombopag or their activators
* Treatment with another investigational product within 30 days or the period 5-fold longer than the half-life of the investigational product, whichever longer, prior to the first dose of eltrombopag
* Prior treatment with eltrombopag, romiplostim, or any other Thrombopoietin (TPO) receptor agonist
* Use of prohibited concomitant medications.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2015-09-10 (Actual); Study Completion 2017-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Japan (9):
  - Novartis Investigative Site, Aichi
  - Novartis Investigative Site, Hyōgo
  - Novartis Investigative Site, Ibaraki
  - Novartis Investigative Site, Ishikawa
  - Novartis Investigative Site, Miyagi
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Tochigi
  - Novartis Investigative Site, Tokyo

REFERENCES:
- [Derived] Yamazaki H, Ohta K, Iida H, Imada K, Obara N, Tokumine Y, Tomiyama Y, Usuki K, Imajo K, Miyamura K, Sasaki O, Fanghong Z, Hattori T, Tajima T, Matsuda A, Nakao S. Hematologic recovery induced by eltrombopag in Japanese patients with aplastic anemia refractory or intolerant to immunosuppressive therapy. Int J Hematol. 2019 Aug;110(2):187-196. doi: 10.1007/s12185-019-02683-1. Epub 2019 Jun 10. PMID 31183813

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place in 12 clinical sites in Japan
Pre-assignment Details: The target number of subjects enrolled was 20. A total 36 subjects were screened and 21 were enrolled in the study. All 21 subjects enrolled received at least 1 dose of study treatment and were included in the planned analysis sets (full analysis set, safety population and pharmacokinetic population).
Period: Overall Study
Arm/Group | Eltrombopag
Started (Full Analysis Set (FAS)) | 21
Safety Set (SS) (All patients who were treated with eltrombopag at least once) | 21
Pharmacokinetic Analysis Set (PAS) (All patients who provided Pharmacokinetics (PK) serum samples) | 21
Completed | 16
Not Completed | 5
Not completed — Investigator discretion | 1
Not completed — Lack of Efficacy | 1
Not completed — Protocol deviation | 1
Not completed — Protocol-defined stopping criteria | 2

BASELINE CHARACTERISTICS:
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: Years] | 53.0 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Hematological Response at Week 26
Description: Hematologic response rate at 6 months (at WeeK 26) after the start of study treatment was defined as the percentage of subjects who met any of the response criteria (Platelet count, Hemoglobin level, Neutrophil count). 1 ) Platelet count: an increase from baseline by 20,000/μL or more (In the absence of platelet transfusion), or no platelet transfusion requirements for 8 weeks; 2) Hemoglobin: When the baseline hemoglobin level is <9 g/dL: Without RBC transfusion at baseline, an increase from baseline by 1.5 g/dL or more; With RBC transfusion at baseline, a decrease of at least 4 units in RBC transfusions in the post-treatment 8-week period compared to the pre-treatment 8-week period (1 unit = RBC derived from 200 mL blood); 3) Neutrophil count: an increase from baseline by 500/μL or more (in the absence of granulocyte colony-stimulating factor (G-CSF)), or (if < 500/μL at baseline) an increase by 100 % or more. Only descriptive analysis done.
Time Frame: D183 (Week 26)
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
Percentage of participants | 47.6 [25.7 to 70.2]

2. Secondary Outcome: Change in Platelet Count From Baseline in the Absence of Platelet Transfusion Over Time
Description: The changes in observed values for Platelet Count were summarized. The measurements were followed up to Week 26 and thereafter in the extension part (Up to the launch of the product after approval, which will be approximately up to two and a half years). Only descriptive analysis done.
Time Frame: Up to 2.5 years
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Mean (Standard Deviation); unit: Giga/Liter (Gi/L)
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
Giga/Liter (Gi/L)
  Baseline | 12.19 (7.155)
  D92 Week13: number analyzed (Participants) | 19
  D92 Week13 | 6.32 (7.698)
  D183 Week26: number analyzed (Participants) | 16
  D183 Week26 | 13.09 (14.015)
  Extension W39: number analyzed (Participants) | 9
  Extension W39 | 23.50 (22.037)
  Extension W52: number analyzed (Participants) | 9
  Extension W52 | 21.50 (15.720)
  Extension W78: number analyzed (Participants) | 8
  Extension W78 | 36.69 (23.798)
  Extension W104: number analyzed (Participants) | 7
  Extension W104 | 35.79 (21.389)
  Extension W130: number analyzed (Participants) | 7
  Extension W130 | 42.79 (28.795)
  Extension W156: number analyzed (Participants) | 1
  Extension W156 | 25.50 (NA) — Not calculated
  Withdrawal: number analyzed (Participants) | 8
  Withdrawal | 8.81 (19.387)
  Last Assessment On-Therapy | 18.38 (24.017)

3. Secondary Outcome: Change in Hemoglobin From Baseline in the Absence of Red Blood Cell (RBC) Transfusion Over Time
Description: The changes in observed values for Hemoglobin were summarized. The measurements were followed up to Week 26 and thereafter in the extension part (Up to the launch of the product after approval, which will be approximately up to two and a half years). Only descriptive analysis done.
Time Frame: Up to 2.5 years
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Mean (Standard Deviation); unit: Gram/Liter (g/L)
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
Gram/Liter (g/L)
  Baseline | 70.4 (13.95)
  D92 Week13: number analyzed (Participants) | 19
  D92 Week13 | 4.9 (11.91)
  D183 Week26: number analyzed (Participants) | 16
  D183 Week26 | 8.8 (17.08)
  Extension W39: number analyzed (Participants) | 9
  Extension W39 | 19.3 (22.29)
  Extension W52: number analyzed (Participants) | 9
  Extension W52 | 24.0 (21.11)
  Extension W78: number analyzed (Participants) | 8
  Extension W78 | 32.8 (19.58)
  Extension W104: number analyzed (Participants) | 7
  Extension W104 | 34.4 (20.44)
  Extension W130: number analyzed (Participants) | 7
  Extension W130 | 31.6 (16.99)
  Extension W156: number analyzed (Participants) | 1
  Extension W156 | 16.0 (NA) — Not calculated
  Withdrawal: number analyzed (Participants) | 8
  Withdrawal | -3.0 (13.85)
  Last Assessment On-Therapy | 10.0 (20.14)

4. Secondary Outcome: Change in Neutrophil Count From Baseline in the Absence of Granulocyte-colony Stimulating Factor (G-CSF) Over Time
Description: The changes in observed values for Neutrophil Count were summarized. The measurements were followed up to Week 26 and thereafter in the extension part (Up to the launch of the product after approval, which will be approximately up to two and a half years). Only descriptive analysis done.
Time Frame: Up to 2.5 years
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Mean (Standard Deviation); unit: Giga/Liter (Gi/L)
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
Giga/Liter (Gi/L)
  Baseline | 0.8247 (0.47985)
  D92 Week13: number analyzed (Participants) | 19
  D92 Week13 | 0.3321 (0.51398)
  D183 Week26: number analyzed (Participants) | 16
  D183 Week26 | 0.2046 (0.43640)
  Extension W39: number analyzed (Participants) | 9
  Extension W39 | 0.4537 (0.87231)
  Extension W52: number analyzed (Participants) | 9
  Extension W52 | 0.5236 (0.58529)
  Extension W78: number analyzed (Participants) | 8
  Extension W78 | 0.8579 (0.62320)
  Extension W104: number analyzed (Participants) | 7
  Extension W104 | 0.6312 (1.05205)
  Extension W130: number analyzed (Participants) | 7
  Extension W130 | 1.1835 (1.97999)
  Extension W156: number analyzed (Participants) | 1
  Extension W156 | -0.1712 (NA) — Not calculated
  Withdrawal: number analyzed (Participants) | 8
  Withdrawal | 0.3246 (0.72222)
  Last Assessment On-Therapy | 0.4307 (1.22084)

5. Secondary Outcome: Hematological Response at Week 13 in Terms of the Platelet Count, Hemoglobin Level and Neutrophil Count
Description: The frequency and percentage were calculated with 95% confidence interval (CI) of responses (which meet each response criteria) of platelet count, hemoglobin and neutrophil count at Week 13.
Time Frame: Week 13
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
Percentage of participants | 61.9 [38.4 to 81.9]

6. Secondary Outcome: Duration of Hematological Response in Participants Who Responded at the Week 13
Description: The duration of haematological response was defined, for subjects who responded at the Week 13 visit, as the number of months from the first date of a response until the first date of a relapse or the date the subject was last assessed. Only subjects with at least 2 response assessments were included in the duration of response assessment. The measurements were followed up to Week 26 and thereafter in the extension part (Up to the launch of the product after approval, which will be approximately up to two and a half years). Only descriptive analysis done.
Time Frame: Up to 2.5 years
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
Months
  Hematological Response: number analyzed (Participants) | 13
  Hematological Response | 10.68 [1.64 to 28.32]
  Platelet/Platelet Transfusion: number analyzed (Participants) | 1
  Platelet/Platelet Transfusion | 32.62 [32.62 to 32.62]
  Hemoglobin/RBC Transfusion Response: number analyzed (Participants) | 8
  Hemoglobin/RBC Transfusion Response | 19.19 [5.54 to 28.37]
  Neutrophils Response: number analyzed (Participants) | 7
  Neutrophils Response | 3.02 [1.64 to 4.63]

7. Secondary Outcome: Volume of (Platelet and RBC) Transfusion in Each Period
Description: The amount of blood transfusion (platelets, RBC) were summarized. The measurements were followed up to Week 26 and thereafter in the extension part (Up to the launch of the product after approval, which will be approximately up to two and a half years). Only descriptive analysis done.
Time Frame: Day 1, Day 92 (Week 13), Day 183 (Week 26), Extension W39 and Extension W52
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
milliliter (mL)
  Day 1 (Platelets): number analyzed (Participants) | 6
  Day 1 (Platelets) | 600.0 (309.84)
  Day 1 (RBC): number analyzed (Participants) | 19
  Day 1 (RBC) | 1663.2 (1083.31)
  Day 92 (Week 13) (Platelets): number analyzed (Participants) | 6
  Day 92 (Week 13) (Platelets) | 400.0 (438.18)
  Day 92 (Week 13) (RBC): number analyzed (Participants) | 17
  Day 92 (Week 13) (RBC) | 1152.9 (978.59)
  Day 183 (Week 26) (Platelets): number analyzed (Participants) | 5
  Day 183 (Week 26) (Platelets) | 280.0 (389.87)
  Day 183 (Week 26) (RBC): number analyzed (Participants) | 14
  Day 183 (Week 26) (RBC) | 800.0 (1131.37)
  Extension W39 (Platelets): number analyzed (Participants) | 2
  Extension W39 (Platelets) | 0.0 (0.00)
  Extension W39 (RBC): number analyzed (Participants) | 8
  Extension W39 (RBC) | 300.0 (848.53)
  Extension W52 (Platelets): number analyzed (Participants) | 2
  Extension W52 (Platelets) | 0.0 (0.00)
  Extension W52 (RBC): number analyzed (Participants) | 8
  Extension W52 (RBC) | 400.0 (1131.37)

8. Secondary Outcome: Frequency of (Platelet and RBC) Transfusion in Each Period
Description: The frequency of blood transfusion (platelets, RBC) were summarized. The measurements were followed up to Week 26 and thereafter in the extension part (Up to the launch of the product after approval, which will be approximately up to two and a half years). Only descriptive analysis done.
Time Frame: Day 1, Day 92 (Week 13), Day 183 (Week 26), Extension W39 and Extension W52
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Mean (Standard Deviation); unit: Tansfusion
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
Tansfusion
  Day 1 (Platelets): number analyzed (Participants) | 6
  Day 1 (Platelets) | 3.0 (1.55)
  Day 1 (RBC): number analyzed (Participants) | 19
  Day 1 (RBC) | 4.1 (2.51)
  Day 92 (Week 13) (Platelets): number analyzed (Participants) | 6
  Day 92 (Week 13) (Platelets) | 2.0 (2.19)
  Day 92 (Week 13) (RBC): number analyzed (Participants) | 17
  Day 92 (Week 13) (RBC) | 2.9 (2.41)
  Day 183 (Week 26) (Platelets): number analyzed (Participants) | 5
  Day 183 (Week 26) (Platelets) | 1.4 (1.95)
  Day 183 (Week 26) (RBC): number analyzed (Participants) | 14
  Day 183 (Week 26) (RBC) | 1.9 (2.64)
  Extension W39 (Platelets): number analyzed (Participants) | 2
  Extension W39 (Platelets) | 0.0 (0.00)
  Extension W39 (RBC): number analyzed (Participants) | 8
  Extension W39 (RBC) | 0.8 (2.12)
  Extension W52 (Platelets): number analyzed (Participants) | 2
  Extension W52 (Platelets) | 0.0 (0.00)
  Extension W52 (RBC): number analyzed (Participants) | 8
  Extension W52 (RBC) | 0.9 (2.47)

9. Secondary Outcome: Percentage of Participants With Reduced Volume of Transfusion (Platelet and RBC)
Description: The proportion of the participants for whom the amount of blood transfusion (platelets and RBC) is decreased was measured and reported as a percentage. The measurements were followed up to Week 26 and thereafter in the extension part (Up to the launch of the product after approval, which will be approximately up to two and a half years). Only descriptive analysis done. This analysis was performed for the subjects who were baseline transfusion dependent.
Time Frame: Up to 2.5 years
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Number; unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
Percentage of participants
  Platelet Transfusion Decrease: number analyzed (Participants) | 5
  Platelet Transfusion Decrease | 83.3
  RBC Transfusion Decrease: number analyzed (Participants) | 14
  RBC Transfusion Decrease | 73.7

10. Secondary Outcome: Percentage of Participants Who Become Transfusion (Platelet and RBC) Independent
Description: The proportion of participants for whom blood transfusion (platelets and RBC) became unnecessary was measured and reported as a percentage. The measurements were followed up to Week 26 and thereafter in the extension part (Up to the launch of the product after approval, which will be approximately up to two and a half years). Only descriptive analysis done. This analysis was performed for the subjects who were baseline transfusion dependent.
Time Frame: Up to 2.5 years
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Number; unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
Percentage of participants
  Platelet Transfusion Independence: number analyzed (Participants) | 6
  Platelet Transfusion Independence | 66.7
  RBC Transfusion Independence: number analyzed (Participants) | 19
  RBC Transfusion Independence | 47.4

11. Secondary Outcome: Long-term Safety and Tolerability of Eltrombopag
Description: The frequency and percentage of subjects who experienced adverse events (AEs), serious adverse events (SAEs) and deaths by primary system organ class (SOC) and MedDRA preferred term were summarized.
Time Frame: Up to 30 days after last dose of study treatment
Population: Safety Analysis Set, all subjects who took at least one dose of study treatment. A subject with multiple adverse events within a primary system organ class was counted only once in the total row. Only descriptive analysis done.
Measure: Number; unit: Percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
Percentage of participants
  AEs by Primary SOC (SOC) | 100
  Grade 1 AEs by Primary SOC (SOC): number analyzed (Participants) | 18
  Grade 1 AEs by Primary SOC (SOC) | 85.7
  Grade 2 AEs by Primary SOC (SOC): number analyzed (Participants) | 17
  Grade 2 AEs by Primary SOC (SOC) | 81.0
  Grade 3 AEs by Primary SOC (SOC): number analyzed (Participants) | 9
  Grade 3 AEs by Primary SOC (SOC) | 42.9
  Grade 4 AEs by Primary SOC (SOC): number analyzed (Participants) | 1
  Grade 4 AEs by Primary SOC (SOC) | 4.8
  Grade 5 AEs by Primary SOC (SOC): number analyzed (Participants) | 0
  SAEs by Primary System Organ Class (SOC): number analyzed (Participants) | 6
  SAEs by Primary System Organ Class (SOC) | 28.6
  Deaths by Primary System Organ Class (SOC): number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With Bleeding Events and Severity of Bleeding
Description: The measurements were followed up to Week 26 and thereafter in the extension part.
Time Frame: Up to 30 days after last dose of study treatment
Population: as for outcome 11
Measure: Number; unit: N° of Participants with Bleeding events
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
N° of Participants with Bleeding events
  AE Bleeding - On Treatment: number analyzed (Participants) | 7
  AE Bleeding - On Treatment | 11
  Grade 1 AE Bleeding - On Treatment: number analyzed (Participants) | 7
  Grade 1 AE Bleeding - On Treatment | 9
  Grade 2 AE Bleeding - On Treatment: number analyzed (Participants) | 2
  Grade 2 AE Bleeding - On Treatment | 2
  AE Bleeding - Followup Phase: number analyzed (Participants) | 1
  AE Bleeding - Followup Phase | 6
  Grade 1 AE Bleeding - Followup Phase: number analyzed (Participants) | 1
  Grade 1 AE Bleeding - Followup Phase | 5
  Grade 2 AE Bleeding - Followup Phase: number analyzed (Participants) | 1
  Grade 2 AE Bleeding - Followup Phase | 1
  SAE Bleeding - On Treatment: number analyzed (Participants) | 7
  SAE Bleeding - On Treatment | 0
  SAE Bleeding - Followup Phase: number analyzed (Participants) | 1
  SAE Bleeding - Followup Phase | 3
  Grade 1 SAE Bleeding - Followup Phase: number analyzed (Participants) | 1
  Grade 1 SAE Bleeding - Followup Phase | 2
  Grade 2 SAE Bleeding - Followup Phase: number analyzed (Participants) | 1
  Grade 2 SAE Bleeding - Followup Phase | 1

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Eltrombopag
Description: At some study sites, full blood sampling for pharmacokinetic (PK) evaluation of Eltrombopag was performed on Day 14 to calculate Cmax, tmax, AUC(0-t), and AUC(0-tau). PK parameters were calculated from plasma concentration-time data using non-compartmental methods.
Time Frame: Day 14 at 25 mg QD (-0.05, 0.15, 0.30, 0.45, 1.00, 1.30 and 24.00), at 50,75 and 100 mg QD (pre-dose)
Population: Pharmacokinetic Analysis Set (PAS), which consisted of all participants with at least one valid PK concentration value, was considered.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
nanogram per milliliter (ng/mL) | 6410 (4200)

14. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) for Eltrombopag
Description: as for outcome 13
Time Frame: Day 14 at 25 mg QD (-0.05, 0.15, 0.30, 0.45, 1.00, 1.30 and 24.00), at 50,75 and 100 mg QD (pre-dose)
Population: as for outcome 13
Measure: Median (Full Range); unit: Hour
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
Hour | 2.00 [1.90 to 7.58]

15. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration Within a Subject Across All Treatments (AUC 0-t) and Over the Dosing Interval (AUC 0-tau) for Eltrombopag
Description: as for outcome 13
Time Frame: Day 14 at 25 mg QD (-0.05, 0.15, 0.30, 0.45, 1.00, 1.30 and 24.00), at 50,75 and 100 mg QD (pre-dose)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Hours*nanograms/milliliter (hr*ng/mL)
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
Hours*nanograms/milliliter (hr*ng/mL)
  AUC(0-t): number analyzed (Participants) | 5
  AUC(0-t) | 123000 (92900)
  AUC(0-tau): number analyzed (Participants) | 3
  AUC(0-tau) | 99200 (119000)

16. Secondary Outcome: Mean Change in Eltrombopag Concentration in Pharmacokinetic Serum Samples Over Time at Days 14 and 15
Description: At every study center, blood samples was be collected on Day 15 of multiple doses of eltrombopag 25 mg to determine the plasma eltrombopag concentration prior to the next dose (trough concentration). In addition, one-point pre-dose blood sampling was performed at every study center on Day 15 of multiple doses of eltrombopag 50 mg, 75 mg and 100 mg to determine trough concentrations. PK parameters were calculated from plasma concentration-time data using non-compartmental methods.
Time Frame: Day 14 (pre-dose, 1, 2, 4, 6, 8 and 24 post-dose), Day 15 (pre-dose)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Eltrombopag
Number analyzed (Participants) | 21
nanogram per milliliter (ng/mL)
  Eltrombopag 25 mg (Day 14) - 0Hr: number analyzed (Participants) | 5
  Eltrombopag 25 mg (Day 14) - 0Hr | 4530 (3870)
  Eltrombopag 25 mg (Day 14) - 1Hr: number analyzed (Participants) | 5
  Eltrombopag 25 mg (Day 14) - 1Hr | 5240 (3740)
  Eltrombopag 25 mg (Day 14) - 2Hr: number analyzed (Participants) | 5
  Eltrombopag 25 mg (Day 14) - 2Hr | 5980 (3990)
  Eltrombopag 25 mg (Day 14) - 4Hr: number analyzed (Participants) | 5
  Eltrombopag 25 mg (Day 14) - 4Hr | 5870 (3870)
  Eltrombopag 25 mg (Day 14) - 6Hr: number analyzed (Participants) | 5
  Eltrombopag 25 mg (Day 14) - 6Hr | 5720 (4130)
  Eltrombopag 25 mg (Day 14) - 8Hr: number analyzed (Participants) | 5
  Eltrombopag 25 mg (Day 14) - 8Hr | 5430 (4170)
  Eltrombopag 25 mg (Day 14) - 24Hr: number analyzed (Participants) | 5
  Eltrombopag 25 mg (Day 14) - 24Hr | 4390 (3680)
  Eltrombopag 25 mg (Day 15) - 0Hr | 3730 (2430)
  Eltrombopag 50 mg (Day 15) - 0Hr: number analyzed (Participants) | 20
  Eltrombopag 50 mg (Day 15) - 0Hr | 8530 (6410)
  Eltrombopag 75 mg (Day 15) - 0Hr: number analyzed (Participants) | 20
  Eltrombopag 75 mg (Day 15) - 0Hr | 15200 (12000)
  Eltrombopag 100 mg (Day 15) - 0Hr: number analyzed (Participants) | 19
  Eltrombopag 100 mg (Day 15) - 0Hr | 19300 (15000)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to approximately 3 years and 1 month.
Arm/Group | Eltrombopag
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 6/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=21)
Retinal detachment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Fibrin D dimer increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=21)
Abdominal pain upper (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Periodontal disease (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Gastroenteritis (Infections and infestations) | 3
Influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 8
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.